CLINICAL TRIAL: NCT03943862
Title: To Share or Not To Share (2Share) - Group Intervention to Support Disclosure Decisions After Suicide Attempt
Brief Title: To Share Or Not To Share
Acronym: 2Share
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to a small number of study participants.
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Nathalie Oexle, Assistant Professor, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 345/18
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: History of Suicide Attempt
Keywords: Stigma; Suicide attempt survivor; Secrecy; Group intervention; Disclosure
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (2Share) + treatment as usual (Experimental): Study participants randomized to the experimental group receive the intervention (2Share) while maintaining their current treatment (treatment as usual). 2Share is a peer-led group intervention containing three two-hour sessions within two weeks plus an additional booster session four weeks later.
  Fidelity to manual is rated in each session by study staff.
  Interventions: Behavioral: 2Share
- Treatment as usual (No Intervention): Participants randomized to the control group do not receive the group program but maintain their current treatment (treatment as usual).

INTERVENTIONS:
Behavioral: 2Share — The peer-led group program contains of three lessons plus one booster session:
  * Lesson 1: Consider the pros and cons of disclosing: Participants reflect on their experience of self-stigma and weigh their pros and cons of (non-)disclosing a suicide attempt.
  * Lesson 2: Different ways to disclose: Participants learn about the different ways to disclose and their respective pros and cons. Afterwards participants develop strategies to choose a person to disclose to, and discuss possible responses they might experience.
  * Lesson 3: Telling your story: Participants learn how to tell their own story.
  * In a booster session, participants will discuss their experiences with disclosure or non-disclosure.
  Arms: Intervention (2Share) + treatment as usual

SUMMARY:
The purpose of the study is to evaluate the group-based intervention "To Share Or Not To Share" in a German clinical setting. Feasibility and efficacy of the program will be tested in a pilot randomized-controlled trial.

DETAILED DESCRIPTION:
People who have survived a suicide attempt often face public and self-stigma, and secrecy is a common strategy to minimize the risk of being labeled. Both secrecy and disclosure have pros and cons. The decision whether, when, and to whom to disclose a previous suicide attempt is complex. Interventions can provide guidance for systematic consideration and a well informed decision. Potentially, it may not be disclosure itself, but the empowered decision for or against disclosure of a previous suicide attempt that reduces distress and leads to beneficial outcomes.

The manualized peer-led group intervention "Honest, Open, Proud" (HOP) supports people with mental illness in their decision whether to disclose mental illness. Research showed positive effects of the intervention on stigma stress, disclosure-related distress and quality of life. Based on HOP, "To Share Or Not To Share" (2Share) was developed to systematically guide suicide attempt survivors through their decision whether and how to disclose a previous suicide attempt.

2Share led to significant reductions in self-stigma and depressive symptoms, as well as increased self-esteem in a recent pilot randomized-controlled trial (RCT) in the US. The aim of the current study is to evaluate 2Share in a German clinical setting. Feasibility and efficacy of 2 Share will be tested in a pilot RCT.

ELIGIBILITY:
Inclusion Criteria:

* Current inpatient, outpatient or day clinical treatment at the Bezirkskrankenhaus Günzburg, Germany
* Age ≥ 18 years
* At least one previous suicide attempt
* Positive screening for disclosure distress (1 item: "In general, how distressed or worried are you in terms of secrecy or disclosure of your suicide attempt?", self-report, persons with a score ≥ 4 on a scale from 1-7 are included)
* Written informed consent
* Sufficient German language skills

Exclusion Criteria:

* Current suicidality (1 item: "Have you had thoughts that you would be better off dead for at least several days during the last week?", self-report, persons responding with yes will be excluded and will be offered support)
* Suicide attempt within the last four weeks
* Dementia or organic disease (ICD-10: F0)
* Primary substance dependence (ICD-10: F1x.2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Self-stigma related to suicide attempt | 2 weeks
  Self-Stigma of Suicide Attempt Survivor Scale (SSSAS), 14-item apply subscale (Sheehan et al, 2018); each item is rated from 1-9, we will calculate a sum score accross all items (range 9-126) with higher scores indicating more self-stigma.

SECONDARY OUTCOMES:
Self-stigma related to suicide attempt | baseline, 6 weeks, 12 weeks
  Self-Stigma of Suicide Attempt Survivor Scale (SSSAS), 14-item apply subscale (Sheehan et al, 2018); each item is rated from 1-9, we will calculate a sum score accross all items (range 9-126) with higher scores indicating more self-stigma.
Self-Stigma (alienation) related to suicide attempt | baseline, 6 weeks, 12 weeks
  Internalized Stigma of Mental Illness scale (ISMI), 6-item alienation subscale (Ritsher et al. 2003) adapted for suicide attempt, 6 items rated from 1-4, we will calculate a mean score accross all items (range: 1-6) with higher scores indicating more self-stigma.
Stigma stress related to suicide attempt | baseline, 2 weeks, 6 weeks, 12 weeks
  Stigma Stress Scale (Rüsch et al., 2009a,b) adapted for suicide attempt, 8-items rated from 1-7 with 4 items measuring the primary appraisal of stigma as harmful and 4 items measuring the secondary appraisal of perceived resources to cope with stigma-related harm, for each of the two subscales we will calculate a mean score (range 1-7) and a total stigma stress score will be caclulated by subtracting perceived resources from perceived harm with higher difference scores (range -6 to +6) indicating more stigma-stress.
Secrecy about suicide attempt | baseline, 2 weeks, 6 weeks, 12 weeks
  Secrecy Scale (Link et al., 1991) adapted for suicide attempt, 5 items rated from 1-6, we will calculate a mean score accross all items (range 1-6) with higher scores indicating more secrecy.
General disclosure distress | baseline, 2 weeks, 6 weeks, 12 weeks
  Distress Disclosure Index (Kahn et al., 2001), 12 items rated from 1-5, we will calculate a sum score accross all items (range 12-60) with higher scores indicating more disclosure distress.
Help-seeking for suicidality | baseline, 2 weeks, 6 weeks, 12 weeks
  General Help-Seeking Questionnaire - suicidal ideation subscale (GHSQ-SI) (Wilson et al., 2005), 10 items rated from 1-7, we will calculate mean scores (range 1-7) for items related to social contacts (items 1-4) and care providers (items 5,7,10).
Depressive symptoms | baseline, 2 weeks, 6 weeks, 12 weeks
  Center for Epidemiological Studies-Depression Scale - short form (CES-D) (Hautzinger et al., 1993), 15 items rated from 0-3, we will calculate a sum score accross all items (range 0-45) with higher scores indicating more depressive symptoms.
Suicidal ideation | baseline, 2 weeks, 6 weeks, 12 weeks
  Suicidal Ideation Attributes Scale (SIDAS) (Spijker et al., 2014), 5 items rated from 0-10, we will calculate a total sum score accross all items (range 0-50) with higher scores indicating more suicidality.
Recovery | baseline, 2 weeks, 6 weeks, 12 weeks
  Recovery Assessment Scale - short version (RAS-G) (Corrigan et al., 2004), 24 items rated from 1-5, we will calculate a mean score accross all items (range 1-5) with higher scores indicating more recovery.
Self-esteem | baseline, 2 weeks, 6 weeks, 12 weeks
  Rosenberg's Self-Esteem Scale (RSE) (Collani et al., 2003), 10 items rated from 0-3, we will caculate a sum score accross all items (range 0-30) with higher scores indicating more self-esteem.
Quality of life | baseline, 2 weeks, 6 weeks, 12 weeks
  EUROHIS Quality of Life Index (EUROHIS-QOL) (Brähler et al., 2007), 8 items rated from 1-5, we will calculate a sum score accross all items (range 8-40) with higher scores indicating more quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ulm and BKH Günzburg, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheehan L, Oexle N, Dubke R, Wan HT, Corrigan PW. The Self-Stigma of Suicide Attempt Survivors. Arch Suicide Res. 2020 Jan-Mar;24(1):34-47. doi: 10.1080/13811118.2018.1510797. Epub 2018 Dec 1. PMID 30142296
- [Background] Rusch N, Corrigan PW, Powell K, Rajah A, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: II. Emotional stress responses, coping behavior and outcome. Schizophr Res. 2009 May;110(1-3):65-71. doi: 10.1016/j.schres.2009.01.005. Epub 2009 Feb 23. PMID 19237266
- [Background] Rusch N, Corrigan PW, Wassel A, Michaels P, Olschewski M, Wilkniss S, Batia K. A stress-coping model of mental illness stigma: I. Predictors of cognitive stress appraisal. Schizophr Res. 2009 May;110(1-3):59-64. doi: 10.1016/j.schres.2009.01.006. Epub 2009 Mar 6. PMID 19269140
- [Background] Link BG, Mirotznik J, Cullen FT. The effectiveness of stigma coping orientations: can negative consequences of mental illness labeling be avoided? J Health Soc Behav. 1991 Sep;32(3):302-20. PMID 1940212
- [Background] Kahn JH, Hessling RM. Measuring the tendency to conceal versus disclose psychological distress. J Soc Clin Psychol. 2001;20(1):41-65. doi:10.1521/jscp.20.1.41.22254
- [Background] Wilson CJ, Deane FP, Ciarrochi JV, Rickwood D. Measuring help seeking intentions: properties of the General Help Seeking Questionnaire. Canadian Journal of Counselling. 2005;39(1):15-28. doi:10.1080/09638237.2017.1370642.
- [Background] Hautzinger M, Bailer M. Allgemeine Depressions-Skala [The German version of the Center for Epidemiological Studies-Depression scale]. Weinheim: Beltz; 1993.
- [Background] van Spijker BA, Batterham PJ, Calear AL, Farrer L, Christensen H, Reynolds J, Kerkhof AJ. The suicidal ideation attributes scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide Life Threat Behav. 2014 Aug;44(4):408-19. doi: 10.1111/sltb.12084. Epub 2014 Feb 24. PMID 24612048
- [Background] Corrigan PW, Salzer M, Ralph RO, Sangster Y, Keck L. Examining the factor structure of the recovery assessment scale. Schizophr Bull. 2004;30(4):1035-41. doi: 10.1093/oxfordjournals.schbul.a007118. PMID 15957202
- [Background] Collani G v., Herzberg PY. Eine revidierte Fassung der deutschsprachigen Skala zum Selbstwertgefühl von Rosenberg [A revision of the German Rosenbergs self-esteem scale]. Zeitschrift für Differentielle und Diagnostische Psychologie. 2003;24(1):3-7. doi:10.1024//0170-1789.24.1.3
- [Background] Brähler E, Mühlan H, Albani C, Schmidt S. Teststatistische Prüfung und Normierung der deutschen Versionen des EUROHIS-QOL Lebensqualität-Index und des WHO-5 Wohlbefindens-Index [Psychometrics and standardization of the German version of EUROHIS-QOL quality of life index and WHO-5 wellbeing index]. Diagnostica. 2007;53(2):83-96. doi:10.1026/0012-1924.53.2.83
- [Background] Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: psychometric properties of a new measure. Psychiatry Res. 2003 Nov 1;121(1):31-49. doi: 10.1016/j.psychres.2003.08.008. PMID 14572622
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617